CLINICAL TRIAL: NCT03651427
Title: Neuroactive Sex Steroids And Their Influence In Glutamatergic Neurotransmission - Effects in Memory and Cognition in Transgender People
Brief Title: Cross-sex Hormone Therapy and Neuronal Plasticity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 150199a
Record Dates: First submitted 2018-08-24; First posted 2018-08-29 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Gender Dysphoria
Keywords: Estradiol;; Brain; glutamate; spectroscopy; hypogonadism
MeSH Terms: conditions — Gender Dysphoria; Hypogonadism | interventions — Estradiol

STUDY DESIGN:
Intervention Model Description: Sel-controlled case series
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transgender Women (Experimental): Transgender women who already completed GAS or that agreed to start gonadotropin release hormone analogue to suppress endogenous sex hormones.
  If the participants were using CSHT in the moment of the study assignment, they were asked to stop hormones for 30 days to evaluate the impact of hypogonadism in the brain.
  After this first assessment, they received prescriptions for Estradiol (equine conjugated oestrogen, or estradiol valerate, or topic 17-beta estradiol formulations) for 60 days, and the impact of CSHT was evaluated again to compare to washout condition.
  Interventions: Drug: Estradiol

INTERVENTIONS:
Drug: Estradiol — Induced hypogonadism and re-institution of CSHT
  Other Names: Drug washout

SUMMARY:
Transgender women (male-to-female) were invited to participate in this study to test the impact of Cross-Sex Hormone Therapy (CSHT) in the brain.

Neuroimaging and cognitive assessment were performed in different time-points to compare the impact of CSHT in the brain.

DETAILED DESCRIPTION:
Sex hormones are known to exert several effect on the brain white matter, cerebral cortex, functional connectivity and neurotransmission. Furthermore, in transgender people, CSHT is know to induce anatomical and functional changes in the brain. However, only a few studies have already been conducted to investigate the effects of sex hormones on the brain accounting for the interference of endogenous gonadal hormones. Also, there is a lack of knowledge about the importance of CSHT after Gender Affirming Surgery (GAS) regarding induced hypogonadism that follows this surgical procedure. Therefore, neuroimaging studies designed to isolate the effect of endogenous gonadal hormones in people with GD urge to be developed.

To fulfil this purpose, transgender women that have already performed GAS and/or were under Gonadotrophin Release Hormone analogues treatment (in order to induce hypogonadism similar to GAS) were invited to interrupt CSHT for at least 30 days to promote sex hormones washout. At the end of the washout, participants performed magnetic resonance imaging, laboratorial analyses for sex hormones and neuro-cognitive assessment. After this first time-point, participants received a new prescription for CSHT containing estradiol (without progesterone) to be used continuously for 60 days, when the same assessments from the end of washout were repeated 60 days after CSHT to compare brain and cognitive longitudinal changes.

At all the time-points, variations in depression scores and anxiety levels were assessed with specific scales.

ELIGIBILITY:
Inclusion Criteria:

* Transgender women
* Age 18 to 60 years old.

Exclusion Criteria:

* Use of psychostimulant drugs
* Use of Antidepressive, Mood Stabiliser, Anti-psychotic, Benzodiazepines, anti-convulsivants, Anorexigenic
* Endocrinological disease (other than diabetes)
* Arterial Hypertensive Disease of Diabetes Mellitus out of control target
* Neurological disease, including stroke or recent cranial trauma with loss or consciousness
* HIV with low CD4 or high viral charge or symptomatic AIDS
* Neoplasia

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-02-13 (Actual); Primary Completion 2019-03-30 (Estimated); Study Completion 2019-03-30 (Estimated)

PRIMARY OUTCOMES:
Glutamate concentration in the left hippocampus | 90 days
  Proton Spectroscopy - magnetic resonance imaging;
  Glutamate concentration in the left hippocampus will be primarily correlated to working memory scores.

SECONDARY OUTCOMES:
Cortical Thickness | 90 days
  Anatomical magnetic resonance imaging
Diffusion track imaging | 90 days
  Micro-Structural magnetic resonance imaging
functional connectivity | 90 days
  functional magnetic resonance imaging
Glutamate concentration in the anterior cingulate cortex and left dorsolateral prefrontal cortex | 90 days
  Proton spectroscopy - magnetic resonance imaging; Glutamate concentration in the left dorsolateral prefrontal cortex will be correlated to over all measures of cognition and executive functioning.
Cognition | 90 days
  Instrument: Wechsler Adult Intelligence Scale (WAIS) version 3. Subscale: Full Scale Intelligence coefficient. Mean: 100 Standard deviation (SD):15 for Brazilian population. Range of classification: 69 and below - Extremely Low 70-79 - Borderline 80-89 - Low Average 90-109 - Average 110-119 - High Average 120-129 - Superior 130 and above - very superior
Operational memory | 90 days
  Subscale from Wechsler Adult Intelligence Scale (WAIS) version 3. Mean: 100 Standard deviation (SD):15 for Brazilian population. 69 and below - Extremely Low 70-79 - Borderline 80-89 - Low Average 90-109 - Average 110-119 - High Average 120-129 - Superior 130 and above - very superior
Verbal memory | 90 days
  Rey Auditory-Verbal Learning Test (RAVLT). Mean and range for Brazilian population:
  1. A1 (Verbal Memory - Immediate recall). Range (in Z-scores): Z <-1.5 are classified as deficit; Z >-1.5 are expected
  2. A5 (Verbal Memory - immediate recall). Range (in Z-scores): Z <-1.5 are classified as deficit; Z >-1.5 are expected
  3. A7 (Verbal Memory - late recall). Range in (Z-scores): Z <-1.5 are classified as deficit; Z >-1.5 are expected
  4. Learning Over Trial (LOT) (Learning capacity). Range (in Z-scores): Z <-1.5 are classified as deficit; Z >-1.5 are expected (please, note the reference for Brazilian population in the section "references" where the mean and standard deviation according to Brazilian population are described for each of the subtest; Salgado et al. (2011).
Language (Verbal Fluency) | 90 days
  Verbal Fluency Tests: (FAS) and Animals.
  Mean and standard deviation (SD) according to age range and years of education:
  Age range for the test: 16-59 years
  Score classification according to years of education:
  1. From 0 to 8 years of education:
     Mean: 38.8 SD: 12.0
  2. From 9 to 12 years of education:
     Mean: 40.5 SD: 10.7
  3. From 12 to 21 years of education:
  Mean: 44.7 SD:11.2
  Range in Z-scores: Z <-1.5 are classified as deficit; Z >-1.5 are expected
Executive function | 90 days
  Stroop Test -Victoria Version.
  Mean and standard deviation (SD) according to the age range and years of education:
  For 19-39 years old + 5-8 years of education:
  Mean: 33.3 SD:11.35
  For 19-39 years old + 9 or more years of education:
  Mean: 41.73 SD: 9.85
  For 40-59 years old + 5-8 years of education:
  Mean: 28 SD: 7.76
  For 40-59 years old + 9 or more years of education:
  Mean: 37.17 SD: 9.98
  Range in Z-scores:
  Z <-1.5 are classified as deficit; Z >-1.5 are expected

CONTACTS AND LOCATIONS:
Overall Officials: Maria Lobato, Dr, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Salgado JV, Malloy-Diniz LF, Abrantes SS, Moreira L, Schlottfeldt CG, Guimaraes W, Freitas DM, Oliveira J, Fuentes D. Applicability of the Rey auditory-verbal learning test to an adult sample in Brazil. Braz J Psychiatry. 2011 Sep;33(3):234-7. doi: 10.1590/s1516-44462011005000007. PMID 21971775
- See also: This references is related to the "verbal memory" evaluation, described in the outcomes. — http://dx.doi.org/10.1590/S1516-44462011005000007